CLINICAL TRIAL: NCT06389747
Title: Effect of Blood Flow Restriction Technique on Pain, Muscle Tone and Strength in Delayed Muscle Soreness
Brief Title: Effect of Blood Flow Restriction Technique on Delayed Onset Muscle Soreness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gamze Aydin, Researcher, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OU
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Pain Intensity
Keywords: pain; muscle strength; muscle tonus
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: participants and assessors will be blind to different intensity BFR groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- %80 BFR group (Active Comparator): %80 intensity BFR technique will be applied to this group.
  Interventions: Other: BFR technique
- %20 BFR group (Active Comparator): %20 intensity BFR technique will be applied to this group.
  Interventions: Other: BFR technique

INTERVENTIONS:
Other: BFR technique — For BFR application, Airbands brand, wireless, automatic training cuffs will be used. During application, it will be ensured that the device module faces forward and the cuff will be fixed in the correct position by wrapping the band around the metal ring. There will be a space between the skin and the cuff that can fit two fingers. The cuff will then be paired via Bluetooth with the Airbands app installed on the phone. BFR cuffs will be placed proximal to the biceps brachii muscle and pressure will be applied. The cuff will be inflated to automatically detect limb pressure. BFR application with 80% pressure to one group of participants and 20% pressure to the other group will be applied simultaneously with the exercise.

SUMMARY:
The aim of our study is to determine and evaluate the effects of blood flow restriction technique on pain, biomechanical properties and strength of the muscle in delayed onset muscle pain in healthy individuals. A Double Blind, Randomized Controlled, prospective study was planned.

DETAILED DESCRIPTION:
All participants will be taken into the DOMS creation protocol. Participants will then be divided into 80% intensity BFR and 20% intensity Blood Flow Restriction technique (BFR) groups and will be included in an exercise protocol accompanied by BFR application.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between the ages of 18-35 (who have not participated in any resistance training program for at least 6 months)

Exclusion Criteria:

* Having a previous musculoskeletal system injury
* Having a condition that prevents resistance exercise
* Having cardiovascular disease
* Using medication for blood pressure control

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-05-28 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | 2 months
  it will be used for assessment of pain intensity, It is scored between 0-10, and higher scores indicate that the situation is getting worse.
myoton | 2 months
  it will be used for assessment of muscle tonus and biomechanic properties, scores are changin according to different parameters.
dynamometer | 2 months
  it will be used for assessment of myscle strength, lower scores indicate that the situation is getting worse.
dolorimeter | 2 months
  it will be used for assessment of pain thresold pressure, lower scores indicate that the situation is getting worse.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Gamze Aydın, Istanbul
  - Istanbul Okan University, Istanbul

IPD SHARING:
Plan to Share IPD: No